CLINICAL TRIAL: NCT04598412
Title: Comparison of Dietary Protein Intake Patterns and Inadequate Protein Intake in Older Adults Among Countries
Status: Completed | Type: Observational
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Collaborators: Hospital General de Occidente (Other)
Responsible Party: Principal Investigator, Juan Ricardo Lopez y Taylor, Director of the Institute of Applied Sciences for Physical Activity and Sport, Centro Universitario de Ciencias de la Salud, Mexico
Other Study IDs: HGO-ICAAFyD18-6
Record Dates: First submitted 2020-10-16; First posted 2020-10-22 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Aging
Keywords: Protein intake; Older adults

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Mexican sample: Aged >60 years (n = 187)
  Interventions: Other: No intervention
- German sample: Aged >75 years (n = 97)
  Interventions: Other: No intervention
- Northamerican sample: Aged >60 years (n = 200)
  Interventions: Other: No intervention
- British sample: Aged >70 years (n = 38)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Cross-sectional

SUMMARY:
The researchers will compare protein intake patterns per day and per meal among older adults from different countries. The analysis will also compare the proportion of inadequate protein intake per day (different cut points), per meal (breakfast, lunch, dinner), and the number of meals per day that reach an adequate protein content.

DETAILED DESCRIPTION:
There will be a literature review in search of other studies reporting protein intake patterns in older adults. These studies must report total, and per-meal protein intake, evaluated through 24-h dietary recalls, food diaries or food frequency questionnaires. Afterwards, the researchers will contact the authors for data requests and analyze the data; these data will also include some demographic variables (e.g. sex, age, height, weight). Once the data are obtained, the patterns of protein intake will be compared among countries with an ANOVA test. As it is very likely that variances and/or sample sizes will be unequal, a Welch's correction and a Dunnett test for post hoc analyses will be performed. This analysis is going to be performed for the whole sample and by sex. Similarly, the proportion of older adults that do not reach the recommended amounts of protein in a daily (0.8, 1.0, 1.2 g/kg/day) and per meal basis (30 g, 0.4 g/kg) will be calculated. These proportions will be compared among countries with a chi-squared test and employing a z-test for proportions (with Bonferroni adjustment) to identify pairwise differences.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling

Exclusion Criteria:

* Incomplete data registries

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community dwelling older adults (>60 y) from different countries.
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2018-08-19 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
Inadequate protein intake per day | One day
  Percentage of older adults that did not eat enough protein per day according to the following cut points: 0.8, 1.0, and 1.2 g/kg/d
Inadequate protein intake per meal | One day
  Percentage of older adults that did not eat enough protein per meal according to the following cut points: 30 g/meal, or 0.4 g/kg/meal
Meals per day with adequate protein content | One day
  The number of meals per day that had enough protein (>30 g/meal, or >0.4 g/kg/meal).

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Gaytán-González, Principal Investigator — University of Guadalajara
Locations (1):
- Instituto de Ciencias Aplicadas a la Actividad Física y al Deporte, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No